CLINICAL TRIAL: NCT03528200
Title: Pilot Study of IV Dyna CT and CBV Imaging Techniques in Preparation for Vascular Embolization Procedures - DYNA EMBOLIZATION
Brief Title: DYNA EMBOLIZATION - Pilot Study of IV Dyna CT and CBV Imaging Techniques
Acronym: DynaEmbo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00043620
Record Dates: First submitted 2015-10-01; First posted 2018-05-17 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Brain Lesions
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dyna Embo (Other): Contrast dye injected through the IV in their arm which helps to see the blood in the arteries using x-ray pictures
  Interventions: Other: Contrast

INTERVENTIONS:
Other: Contrast — The scan requires that the patient lie still on a hard surface for about 5-10 minutes. Before the scan, they will have a special fluid called contrast dye injected through the IV in their arm. This contrast dye helps to see the blood in the arteries using x-ray pictures.
  After the IV dyna CBV is completed, they will have their routine conventional angiography to evaluate the lesion for embolizable arteries as part of routine clinical care. If the patient undergoes embolization of the lesion (as part of the standard of care), a post embolization Dyna CBV will be performed.
  Other Names: iodinated contrast

SUMMARY:
This is a prospective pilot study evaluating the efficacy of DynaCT in direct comparison to conventional catheter angiography in demonstrating the anatomic details of the vessels supplying brain lesions. Forty patients will be recruited for this pilot study.

DETAILED DESCRIPTION:
There are common intracranial lesions that have increased vascularity that makes surgical resection difficult. Embolization can improve the surgical procedure by easing the resection, decreasing blood loss during surgical resection, and improving visibility of the surgical bed during resection. Conventional intra-arterial (IA) angiography is the gold standard to evaluating pathologies for embolization candidates, however the invasiveness of the procedure (with associated risks), time requirements, and resource utilization of evaluating and possibly embolization of these patients are precluding its widespread use.

Devising a test methodology that is quick, with less risk, and can accurately detect arteries that are of value in embolizing these pathologies will improve the utilization as a screening tool and will result in improved resource utilization that focuses only on those patients that require embolization. Lastly, by correlating the Dyna CBV to surgical resection quality (ease of resection, blood loss from surgical site), a non-invasive, controlled method to evaluating embolization quality can be established to aid surgeons in pre-operative planning as well as serve as a method of evaluating embolization materials designed for the blood vessels associated with brain lesions.

The DynaCT technique is a fully FDA-approved application of the Siemens imaging system and software. DynaCT is often performed during our angiographic and interventional procedures. Neurointerventionists have begun to apply this technology within their practices, and the investigators have selectively applied DynaCT for various clinical applications. However, at this point the investigators have not incorporated the technology into clinical care for patients with intracranial lesions.

Although DynaCT is an approved technology, there have been recent improvements in the software performing the 3D reconstruction. These new features will be used in this study and thus the investigators consider them to be "research scans."

Study patients will provide informed consent for the scan and the patients will not be billed for the DynaCT portion of the procedure (only the standard of care conventional angiography). The investigators have specifically chosen to image patients already undergoing conventional angiography for surgical resection in order to have a direct comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to have an intracranial lesion evaluated for possible surgical resection.

Exclusion Criteria:

1. Patients with severe contrast allergies
2. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
CBV Comparison | One week
  Compare a baseline IV Dyna CBV pre-embolization and immediate post embolization CBV to assess quality of vascular embolization.
Correlation of CBV | One week
  Correlate changes in CBV (post embolization to pre-embolization, and CBV in patients who did not get embolization) to improved surgical procedure (ease of resection, surgical blood loss).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States